CLINICAL TRIAL: NCT00877253
Title: Open-label, Multicenter, Phase I Trial to Evaluate Efficacy and Safety of the Combination Therapy of Genexol®-PM Plus Carboplatin as a Firstline Treatment in Subjects With Advanced Ovarian Cancer
Brief Title: Determine MTD, Evaluate Efficacy and Safety of Genexol®-PM Plus Carboplatin With Advanced Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPMOC201
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — genexol-PM

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose Level One (Experimental)
  Interventions: Drug: Genexol-PM 220mg/㎡, Carboplatin 5AUC
- Dose Level Two (Experimental)
  Interventions: Drug: Genexol-PM 260mg/㎡, Carboplatin 5AUC
- Dose Level Three (Experimental)
  Interventions: Drug: Genexol-PM 300mg/㎡, Carboplatin 5AUC

INTERVENTIONS:
Drug: Genexol-PM 220mg/㎡, Carboplatin 5AUC — Genexol-PM 220mg/m2 by IV infusion over 3 hours on day 1 of every 21 day cycle. Carboplatin, AUC 5 given by IV infusion over 30-60 minutes on day 1 of every 21 day cycle.
  Arms: Dose Level One
Drug: Genexol-PM 260mg/㎡, Carboplatin 5AUC — Genexol-PM 260mg/m2 by IV infusion over 3 hours on day 1 of every 21 day cycle. Carboplatin, AUC 5 given by IV infusion over 30-60 minutes on day 1 of every 21 day cycle.
  Arms: Dose Level Two
Drug: Genexol-PM 300mg/㎡, Carboplatin 5AUC — Genexol-PM 300mg/m2 by IV infusion over 3 hours on day 1 of every 21 day cycle. Carboplatin, AUC 5 given by IV infusion over 30-60 minutes on day 1 of every 21 day cycle.
  Arms: Dose Level Three

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of Genexol®-PM plus Carboplatin and evaluate the efficacy and safety of Genexol®-PM plus Carboplatin regimen in subjects with advanced ovarian cancer.

DETAILED DESCRIPTION:
This is a phase I trial to determine the maximum tolerated dose and recommended phase II dose of the combination therapy with Genexol®-PM and Carboplatin and to evaluate the efficacy and safety of Genexol®-PM when administered with Carboplatin in subjects with advanced ovarian cancer after debulking surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years old.
* Signed informed consent before inclusion.
* Subjects who have histologically or cytologically confirmed advanced epithelial ovarian cancer.(FIGO IIIB-IV)
* Subjects who have measurable disease by RECIST after debulking surgery.
* ECOG performance status of 0, 1, or 2.
* Estimated life expectancy of more than 6 months
* Subjects who have the clinically acceptable function of blood, kidney and liver at screening visit

  * Hb ≥ 10g/dl
  * ANC ≥ 1.5×10^9/L
  * Platelet Count ≥ 100×10^9/L
  * Serum total bilirubin ≤ 1.5×ULN
  * Serum AST and ALT ≤ 2.5×ULN
  * Serum ALP ≤ 2.5×ULN
  * Serum creatinine ≤ 1.5×ULN

Exclusion Criteria:

* Subjects who have received chemotherapy for ovarian cancer other than debulking surgery.
* Subjects who have a history of radiotherapy to pelvis or abdominal cavity
* Subjects who receive immunotherapy or hormonal therapy for ovarian cancer
* Subjects who have other malignancies within the past 5 years
* Subjects who have had a major surgery other than debulking surgery within 2 weeks prior to the screening/baseline visit
* Subjects who have a history of metastasis or currently have a metastasis to the central nervous system(CNS)
* Subjects who have a preexisting sensory or motor neuropathy of grade ≥ 1 based on NCI CTCAE V3.0
* Subjects who have serious medical condition

  * Uncontrolled or severe cardiovascular disease(Ischemic heart disease, myocardial infarction within the last 6 months, congestive heart failure)
  * Uncontrollable infection
  * Previous allergic reactions in connection with paclitaxel and carboplatin
* Subjects who participate another clinical trial within the last 4 weeks before inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Determine the MTD and recommended phase II dose of the combination therapy with Genexol-PM and Carboplatin in subjects with advanced ovarian cancer. | until either MTD is achieved or maximum planned dose is tested

SECONDARY OUTCOMES:
Objective Response Rate (Complete Response (CR) + Partial Response (PR)) | about 1 year (until end of trial)
Time to Tumor Progression | about 1 year (until end of trial)
Overall Survival | about 1 year (until end of trial)
Safety profiles | about 1 year (till end of trial)

CONTACTS AND LOCATIONS:
Overall Officials: Soon Beom Kang, MD, PhD, Principal Investigator — Seoul National University Hospital; Yong Man Kim, MD, PhD, Principal Investigator — Asan Medical Center; Byoung Gie Kim, MD, PhD, Principal Investigator — Samsung Medical Center; Young Tae Kim, MD, PhD, Principal Investigator — Yonsei University Health System Severance Hospital